CLINICAL TRIAL: NCT04343872
Title: UAB Diabetes Research Center (DRC): Chronic Disease and the Reduction of Health Disparities Supplement
Brief Title: Preventing Diabetes in the Deep South: Extending Partnerships and Adapting Interventions to Reach Rural Communities at High Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Cherrington, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300005012; 3P30DK079626-12S1 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Pre-diabetes
Keywords: Obesity; Metformin Therapy
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive lifestyle modification alone (DPP) (Active Comparator): Participants in this arm will receive a lifestyle modification intervention program facilitated by Peer Coach (PC) services
  Interventions: Behavioral: Receive lifestyle modification alone
- Receive lifestyle modification with metformin therapy (Experimental): Participants in this arm will receive a lifestyle modification intervention program facilitated by Peer Coach (PC) services plus metformin recommendation
  Interventions: Behavioral: Receive lifestyle modification alone; Behavioral: Metformin therapy

INTERVENTIONS:
Behavioral: Receive lifestyle modification alone — Participants will receive a 12-month lifestyle intervention program (telehealth + peer coach). The intervention comprises of the Center for Disease Control and Prevention (CDC)-adapted DPP Prevent Type 2 (PreventT2) lifestyle intervention program consisting of 26 classes delivered by trained health educators via telehealth. Additionally, the peer coach provides ongoing support over 12-months with tapered calls mirroring ongoing classes. Participants are randomized at the practice level. Two clinics will be randomized to receive the lifestyle intervention program alone.
Behavioral: Metformin therapy — The two other clinics will be randomized to receive the lifestyle intervention program (described above) with METFORMIN therapy recommendations. Participants are randomized at the practice level. The primary care provider at the clinic will prescribe metformin and participants would be encouraged to take it if the primary care provider consider prescribing.
  Arms: Receive lifestyle modification with metformin therapy

SUMMARY:
Diabetes is responsible for a huge and growing burden of patient suffering and social costs, and the impact of this disease is shared disproportionately by minorities and in rural resource-challenged communities, particularly in the Deep South. To address this problem, the University of Alabama (UAB) Diabetes Research Center (DRC) will establish a primary care clinical network in rural counties of Alabama and in the Mississippi delta that will provide the (DRC) and its members with opportunities for partnership and the infrastructure to conduct translational and clinical research in those patients with the greatest need. A pilot trial will be conducted within the coalition to assess feasibility for a larger trial to evaluate a novel and sustainable approach for diabetes prevention that involves an innovative lifestyle intervention combined with metformin.

DETAILED DESCRIPTION:
The pilot trial in aim three will include enrolling four primary care practices. Each of the participating practices will be randomized to one of two arms and accordingly enrolled participants from each clinic will be assigned to one of two conditions:

Condition 1. Receive lifestyle modification alone (Diabetes Prevention Program (DPP).

Condition 2. Receive lifestyle modification (DPP) with metformin therapy recommendation.

Twenty five participants will be enrolled from each participating practice. Participants will be followed up for 12-14 months after recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 65 years
* Body mass index (BMI) ≥30
* Receives care at one of the participating primary care clinics
* HbA1c 6.0% to 6.4%
* Resides in one location at least 5 days each week
* Willing to attend group-based classes
* Willing to work with a peer advisor in-person and over the phone
* Has regular access to telephone or cellular phone
* Willing and able to use telemonitoring body weight to conduct daily self-weighing
* Estimated Glomerular Filtration Rate (eGFR) of ≥60 in their medical record within 6 months

Exclusion Criteria:

* Diabetes diagnosis or HbA1c >6.4% or fasting glucose ≥126
* HbA1c <6.0%
* Pregnancy or anticipating pregnancy
* Unwilling or unable to do any of the following: give informed consent, accept random assignment, allow study staff to visit them at their primary care clinic for two follow-up visits
* Likely to relocate within next 6 months and no longer be seen at clinic within the next 12 months
* Weight loss ≥5% of body weight in past 6 months (other than postpartum)
* Past bariatric surgery
* Prescription weight loss medications within the past 6 months
* eGFR < 60 within past 6 months
* Unable to ambulate
* Have end-stage medical conditions with limited life expectancy

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cherrington, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinic
Period: Overall Study
Arm/Group | Receive Lifestyle Modification Alone (DPP) | Receive Lifestyle Modification With Metformin Therapy
Started | 29; 2 Clinic | 7; 2 Clinic
Completed | 23; 2 Clinic | 4; 2 Clinic
Not Completed | 6; 0 Clinic | 3; 0 Clinic
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receive Lifestyle Modification Alone (DPP) | Receive Lifestyle Modification With Metformin Therapy | Total
Number analyzed (Participants) | 29 | 7 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 7 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (10.3) | 47.0 (12.3) | 49.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 6 | 30
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 5 | 25
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 7 | 36
Body Weight [Mean (Standard Deviation); unit: pounds] | 264.4 (44.78) | 251.9 (69.07) | 258.3 (57.27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Change in body weight from baseline to 12-months
Time Frame: 12 months
Population: Participants lost to follow-up
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Receive Lifestyle Modification Alone (DPP) | Receive Lifestyle Modification With Metformin Therapy
Number analyzed (Participants) | 23 | 4
Pounds | -3.6 (11.87) | -4.4 (3.21)

2. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in glycosylated hemoglobin (HbA1c) point of care test values
Time Frame: 12 months
Population: Participants lost to follow-up
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Receive Lifestyle Modification Alone (DPP) | Receive Lifestyle Modification With Metformin Therapy
Number analyzed (Participants) | 23 | 4
Percentage of glycosylated hemoglobin | -0.1 (0.52) | -0.5 (0.99)

ADVERSE EVENTS:
Time Frame: 12-months
Arm/Group | Receive Lifestyle Modification Alone (DPP) | Receive Lifestyle Modification With Metformin Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/7
Other Adverse Events (participants affected / at risk) | 0/29 | 0/7

LIMITATIONS AND CAVEATS:
COVID-19 greatly impacted ability to recruit participants and retain participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT04343872/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT04343872/ICF_001.pdf